CLINICAL TRIAL: NCT00291733
Title: Levetiracetam Administration for the Management of Levodopa-Induced Dyskinesias in Parkinson's Disease: A Double-Blind,Placebo-Controlled, Crossover Trial
Brief Title: Levetiracetam Administration for the Management of Levodopa-Induced Dyskinesias in Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: 1st Hospital of Social Security Services (Other)
Collaborators: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VALID-PD
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Levodopa Induced Dyskinesia
Keywords: Levetiracetam; Levodopa-induced dyskinesias; Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Active Comparator): 500mg levetiracetam for one week and 1000mg levetiracetam for one week
  Interventions: Drug: Levetiracetam
- 2 (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- 3 (Active Comparator): After crossover arm 3 equals arm 1
  Interventions: Drug: Levetiracetam
- 4 (Placebo Comparator): After crossover arm 4 equals arm 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — 500mg (2 tabl of 250) for one week and 1000mg (4 tabl of 250) for one week
  Arms: 1; 3
Drug: Placebo — Placebo tabl
  Arms: 2; 4

SUMMARY:
Levodopa-induced dyskinesias have been associated with irregular oscillatory discharge characteristics of basal ganglia. From the other hand, LEV which shares a different electrophysiologic profile than other antiepileptics, inhibits hyper-synchronization of abnormal neuronal firing in experimental models of epilepsy. LEV also reduces levodopa-induced dyskinesias in MPTP-lesioned macaques and modulates "priming phenomenon" which associated with long-term changes in synaptic function that can lead to dyskinesias in PD.

Study objectives :

* To evaluate the effects of levetiracetam (LEV) in two doses (500 and 1000mg) vs placebo on disabling dyskinesias that develop as result of long-term treatment with levodopa, occurring at the time of maximal clinical improvement in patients with Parkinson's disease (PD).
* To evaluate the safety of LEV in patients with PD and antiparkinsonian medication.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of PD will be according to the criteria of United Kingdom Parkinson's Disease Society Brain Bank.

Other inclusion criteria:

* Patients between ages 30 and 80
* Hoehn and Yahr stage of PD over IIb
* Levodopa-induced dyskinesias (LID) despite optimization of antiparkinsonian medication
* LID severity 2 on item 32 and duration 2 on item 33 of the Unified Parkinson's Disease Rating Scale (UPDRS) part IV
* Patient is willing to adhere to protocol requirements as evidence by written informed consent

Exclusion Criteria:

* Patient has a history of any medical condition or clinically significant laboratory abnormalities that can subject them to unwarranted risk.
* Female patient is pregnant or breastfeeding or has not been using or was not continuing to use an adequate contraceptive method for the last 30 days, or is not at least one year post-menopausal.
* Patient with ablative surgeries or DBS implantation electrodes for diseases of the basal ganglia.
* Patient has a low Mini-mental Examination MMSE score <25 or has a history of bipolar psychosis or schizophrenia.
* Patient is unwilling to sign an informed consent or to comply with protocol requirements.
* Patient is taking or has taken in the past month amantadine.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-05; Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Percent change of "on with levodopa-induced dyskinesias (LID)" time from patient diaries | 24 hours

SECONDARY OUTCOMES:
Percent change of "on without dyskinesias" and "off" time from patient diaries. Changes in severity and duration of LID according to the UPDRS , Schwab & England scale and also Goetz dyskinesia scale after a levodopa challenge dose. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pantelis Stathis, MD, Study Chair — 1st Hospital of Social Security Services; Spiros Konitsiotis, MD, Principal Investigator — Department of Neurology, University of Ioannina; Vasilis Kyriakakis, MD, Principal Investigator — Department of Neurology, General Hospital of Lamia; Georgios Tagaris, MD, Principal Investigator — Department of Neurology, PGNA "Georgios Genimatas"; Kostas Papadopoulos, MD, Principal Investigator — Department of Neurology, Hospital of Mental Diseases of Tripolis
Locations (1):
- Department of Neurology, 1st Hospital of Social Security Services, Athens, Greece